CLINICAL TRIAL: NCT02580955
Title: ReFlow Study, a Physician-initiated Trial Investigating the Efficacy of the LegFlow Paclitaxel-Eluting Peripheral Balloon Dilatation Catheter for the Treatment of Femoropopliteal Lesions Longer Than 15cm (TASC C&D Lesions).
Brief Title: REFLOW Study, Investigating the Efficacy of the LEGFLOW DCB in TASC C&D Fempop Lesions
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-150527
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEGFLOW DCB (Experimental): patients treated with the LEGFLOW Paclitaxel-Eluting Peripheral Balloon Dilatation Catheter
  Interventions: Device: LEGFLOW DCB

INTERVENTIONS:
Device: LEGFLOW DCB

SUMMARY:
A physician initiated trial investigating the LEGFLOW Paclitaxel-Eluting Peripheral Balloon dilatation catheter for the treatment of femoropopliteal lesions longer than 15cm.

Objective: to evaluate the short-term outcome of the treatment by means of the LEGFLOW Paclitaxel-Eluting Peripheral BAlloon Dilattaion for the treatment of long femoropopliteal lesions (TASC C&D).

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting a score from 2 to 5 following Rutherford classification
2. Patient is willing to comply with specified follow-up evaluations at the specified times
3. Patient is >18 years old
4. Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
5. Patient has a projected life expectancy of at least 12 months
6. Prior to enrolment, the guidewire has crossed target lesion
7. Patient is eligible for treatment with the LEGFLOW Paclitaxel-Eluting Peripheral Balloon Dilatation Catheter
8. Male, infertile female or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure
9. De novo lesion located in the femoropopliteal arteries suitable for endovascular therapy
10. The target lesion is located within the native femoropopliteal artery
11. The length of the target lesion is > 150mm and considered as TASC C or D lesion according to the TASC II classification.
12. The target lesion has angiographic evidence of stenosis > 50% or occlusion which can be passed with standard guidewire manipulation
13. Target vessel diameter visually estimated is >4mm and <6.5 mm
14. There is angiographic evidence of at least one-vessel-runoff to the foot, irrespective of whether or not outflow was re-established by means of previous endovascular intervention

Exclusion Criteria:

1. Patient refusing treatment
2. Presence of a stent in the target lesion that was placed during a previous procedure
3. Untreated flow-limiting inflow lesions
4. Any previous surgery in the target vessel (including prior ipsilateral crural bypass)
5. Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
6. Previous bypass surgery in the same limb
7. Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
8. Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
9. Perforation at the angioplasty site evidenced by extravasation of contrast medium
10. Patients with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
11. Patients with uncorrected bleeding disorders
12. Aneurysm located at the level of the SFA
13. Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
14. Severe medical comorbidities (untreated CAD/CHF, sever COPD, metastatic malignancy, dementia, etc.) or other medical condition that would preclude compliance with the study protocol or 1-year life expectancy
15. Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
16. Septicemia or bacteremia
17. Ipsilateral iliac treatment before the target lesion procedure with a residual stenosis >30% or ipsilateral iliac treatment conducted after the target lesion procedure
18. Use of thrombectomy, atherectomy or laser devices during procedure
19. Any patient considered to be hemodynamically unstable at onset of procedure
20. Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
21. Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Primary Patency at 12 months, defined as absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) at the target lesion and without TLR within 12 months. | 12 months

SECONDARY OUTCOMES:
Primary Patency rate at 1 & 6 month follow-up | 1 month, 6 months
Technical success | during procedure, at baseline
Freedom from TLR at 1,6 and 12-month follow-up | 1 month, 6 months, 12 months
Clinical success at follow-up, defined as an improvement of Rutherford classification at all follow-up time points | 12 months
Serious adverse events | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - OLV Hospital, Aalst
  - Imelda Hospital Bonheiden, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - Heilig Hart Hospital, Tienen